CLINICAL TRIAL: NCT03554083
Title: Neoadjuvant Therapy for Patients With High Risk Stage III Melanoma: A Pilot Clinical Trial
Brief Title: Vemurafenib, Cobimetinib, Atezolizumab, and Tiragolumab in Treating Patients With High-Risk Stage III Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1776; NCI-2018-01018 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1776 (Other: Mayo Clinic in Rochester); 17-009383 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8
MeSH Terms: interventions — atezolizumab; cobimetinib; Tiragolumab; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A - CLOSED (vemurafenib, cobimetinib, atezolizumab) (Experimental): Patients receive vemurafenib PO BID on days 1-28 and cobimetinib PO QD on days 1-21. Patients also receive atezolizumab intravenously (IV) over 30-60 minutes on days 1 and 15 of cycles 2 and 3. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Within 2-4 weeks after treatment, patients undergo surgery then receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Vemurafenib
- Arm B - CLOSED (cobimetinib, atezolizumab) (Experimental): Patients receive cobimetinib as in Arm A and atezolizumab IV over 30-60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Within 2-4 weeks after treatment, patients undergo surgery then receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- Arm C (atezolizumab, tiragolumab) (Experimental): Patients with BRAF wild-type or BRAF mutant melanoma receive atezolizumab IV over 30-60 minutes and tiragolumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Biological: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518
  Arms: Arm A - CLOSED (vemurafenib, cobimetinib, atezolizumab); Arm B - CLOSED (cobimetinib, atezolizumab)
Biological: Tiragolumab — Given IV
  Other Names: MTIG7192A; RG6058
  Arms: Arm C (atezolizumab, tiragolumab)
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX-4032; PLX4032; RG 7204; RG7204; RO 5185426; Zelboraf
  Arms: Arm A - CLOSED (vemurafenib, cobimetinib, atezolizumab)

SUMMARY:
This trial studies how well vemurafenib, cobimetinib, and atezolizumab work in treating patients with high-risk stage III melanoma. Vemurafenib and cobimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as atezolizumab and tiragolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving vemurafenib, cobimetinib, and atezolizumab may work better in treating high-risk stage III melanoma. Giving atezolizumab and tiragolumab together may also work better in treating high-risk stage III melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the percentage of patients with stage III BRAFV600 mutated (BRAFm) melanoma that achieves a pathologic complete response after 12 weeks of neoadjuvant vemurafenib/cobimetinib/atezolizumab (neoadjuvant phase).

II. To estimate the percentage of patients with stage III BRAF-wild-type (BRAFwt) melanoma that achieves a pathologic complete response after 12 weeks of neoadjuvant cobimetinib/atezolizumab (neoadjuvant phase).

III. To estimate the percentage of patients with stage III melanoma that achieves a pathologic complete response (pCR) after 12 weeks of neoadjuvant atezolizumab/tiragolumab (neoadjuvant phase).

IV. To assess recurrence-free survival (RFS) in patients with stage III BRAFm melanoma after neoadjuvant vemurafenib/cobimetinib/ atezolizumab, surgery, and adjuvant atezolizumab (adjuvant phase).

V. To assess RFS in patients with stage III BRAFwt melanoma after neoadjuvant cobimetinib/atezolizumab, surgery, and adjuvant atezolizumab (adjuvant phase).

VI. To assess RFS in patients with stage III melanoma after neoadjuvant atezolizumab/tiragolumab, surgery, and adjuvant atezolizumab (adjuvant phase).

SECONDARY OBJECTIVES:

I. To determine the frequency of adverse events among patients with stage III BRAFm melanoma receiving neoadjuvant vemurafenib / cobimetinib / atezolizumab followed by surgery followed by adjuvant atezolizumab.

II. To determine the frequency of adverse events among patients with stage III BRAFwt melanoma receiving neoadjuvant cobimetinib/atezolizumab followed by surgery followed by adjuvant atezolizumab.

III. To determine the frequency of adverse events among patients with stage III melanoma receiving neoadjuvant atezolizumab/tiragolumab followed by surgery followed by adjuvant atezolizumab.

TRANSLATIONAL OBJECTIVES:

I. To determine the association between pretreatment, on treatment, post-neoadjuvant and post-adjuvant treatment soluble PD-L1 (sPD-L1) and RFS in patients with stage III melanoma receiving neoadjuvant vemurafenib / cobimetinib / atezolizumab or cobimetinib/atezolizumab, or atezolizumab/tiragolumab, followed by surgery and adjuvant atezolizumab.

II. To determine the association between pretreatment, on treatment, post-neoadjuvant and post-adjuvant treatment intracellular bim in tumor-related T cells and RFS in patients with stage III melanoma after neoadjuvant vemurafenib/cobimetinib/atezolizumab or cobimetinib/atezolizumab, or atezolizumab/tiragolumab, followed by surgery and adjuvant atezolizumab.

III. Evaluate associations between pre and post-neoadjuvant treatment molecular features of melanomas and the tumor immune microenvironment in responders versus non-responders with multiplex immunofluorescence (MxIF) (including T-cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine-based inhibition motif domains [TIGIT]) and ribonucleic acid-sequencing (RNA-Seq) in patients with stage III melanoma after neoadjuvant vemurafenib/cobimetinib/atezolizumab or cobimetinib/atezolizumab, or atezolizumab/tiragolumab, followed by surgery and adjuvant atezolizumab.

IV. To determine the association between pretreatment tumor PD-L1, pCR, and RFS in patients with stage III melanoma receiving neoadjuvant vemurafenib/ cobimetinib/ atezolizumab or cobimetinib/atezolizumab, or atezolizumab/tiragolumab, followed by surgery and adjuvant atezolizumab.

V. To evaluate changes in cell-free deoxyribonucleic acid (DNA) over time to determine whether these changes correlate with clinical outcomes, including pathologic complete response and cancer progression.

VI. To compare T cell receptor diversity/clonality in pretreatment tumor, tumor and uninvolved lymph node from the time of surgery, as well as blood from before treatment, after neoadjuvant treatment, after surgery, and after adjuvant treatment.

VII. To compare the frequency of neoantigen-specific T cells in pretreatment tumor, tumor and uninvolved lymph node from the time of surgery, as well as blood from before treatment, after neoadjuvant treatment, after surgery, and after adjuvant treatment.

VIII. To compare peripheral blood mononuclear cell subsets from before treatment, after neoadjuvant treatment, after surgery, and after adjuvant treatment via multiparametric mass cytometry (CyTOF).

IX. To assess whether treatment response to neoadjuvant systemic therapy in the index biopsy-proven metastatic node is indicative of the overall response in the nodal basin.

X. To evaluate whether baseline or changes over time in microbiome samples correlate with clinical outcomes, including pathologic complete response and cancer progression.

OUTLINE: Patients are assigned to Arm C.

ARM A (BRAF mutant): Patients receive vemurafenib orally (PO) twice daily (BID) on days 1-28 and cobimetinib PO once daily (QD) on days 1-21. Patients also receive atezolizumab intravenously (IV) over 30-60 minutes on days 1 and 15 of cycles 2 and 3. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. (CLOSED TO ACCRUAL)

ARM B (BRAF wild-type): Patients receive cobimetinib as in Arm A and atezolizumab IV over 30-60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. (CLOSED TO ACCRUAL)

ARM C: Patients with BRAF wild-type or BRAF mutant melanoma receive atezolizumab IV over 30-60 minutes and tiragolumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

Within 2-4 weeks after treatment, patients undergo surgery then receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Age >= 18 years
* PRE-REGISTRATION: High-risk stage III melanoma, defined as (any of the following):

  * Recurrent nodal metastasis, or
  * Clinically detectable nodal metastasis, or
  * Metastatic involvement of more than one nodal basin
  * NOTE: For the purpose of pre-registration, high-risk stage III melanoma is defined based on clinical and imaging assessment (positron emission tomography/computed tomography [PET/CT], CT, or magnetic resonance imaging [MRI]). Histologic confirmation of nodal metastatic disease is not needed at the time of pre-registration, provided there is histologic confirmation of primary melanoma or a prior lymph node metastasis.
* PRE-REGISTRATION: Willing to submit archival tissue from a lymph node biopsy or undergo a needle biopsy (with clip placement) for BRAF testing and for research purposes.
* PRE-REGISTRATION: Willing to forego anticancer treatments or investigational agents during pre-registration period.
* PRE-REGISTRATION: The following laboratory values obtained =< 28 days prior to pre-registration:

  * Only for patients receiving therapeutic anticoagulation: stable anticoagulant regimen and stable international normalized ratio (INR).
* REGISTRATION: Histologic confirmation of stage III melanoma, as defined by the American Joint Committee on Cancer, 8th revised edition.
* REGISTRATION: Arms A and B only: Documentation of BRAFV600 mutation status in melanoma tumor tissue (archival or newly obtained) through use of a Clinical Laboratory Improvement Amendments (CLIA)-approved clinical mutation test.
* REGISTRATION: Surgically resectable disease, as determined by a melanoma surgical oncologist.
* REGISTRATION: Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* REGISTRATION: Life expectancy >= 26 weeks.
* REGISTRATION: Absolute neutrophil count (ANC) >= 1500/mm^3 obtained =< 14 days prior to registration.
* REGISTRATION: Platelet count >= 100,000/mm^3 obtained =< 14 days prior to registration.
* REGISTRATION: Hemoglobin >= 9.0 g/dL obtained =< 14 days prior to registration.
* REGISTRATION: Direct bilirubin =< institutional upper limit of normal (ULN) obtained =< 14 days prior to registration.
* REGISTRATION: Aspartate transaminase (AST) and alanine transaminase (ALT) =< 2 x ULN obtained =< 14 days prior to registration.
* REGISTRATION: Alkaline phosphatase < 2.5 x ULN obtained =< 14 days prior to registration.
* REGISTRATION: Creatinine =< 1.5 x ULN or creatinine clearance (CrCl) >= 45 mL/min on the basis of measured CrCl from a 24-hour urine collection or Cockcroft-Gault glomerular filtration rate estimation obtained =< 14 days prior to registration.
* REGISTRATION: Arms A and B only: Left ventricular ejection fraction (LVEF) >= 50% or institutional lower limit of normal (LLN) =< 6 months prior to registration.
* REGISTRATION: Arms A and B only: Average corrected QT interval (QTc) =< 450 ms on triplicate 12 lead electrocardiography (ECG) =< 28 days prior to registration.

  * NOTE: QTc intervals will be corrected using Fridericia's formula.
* REGISTRATION: Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only.
* REGISTRATION: For persons of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for 6 months after the last dose of study treatment.
* REGISTRATION: For persons able to father a child: agreement to remain abstinent (refrain from heterosexual intercourse with a person of childbearing potential) or use contraceptive measures, and agreement to refrain from donating sperm during the treatment period and for 6 months after the last dose of study treatment.
* REGISTRATION: Provide written informed consent.
* REGISTRATION: Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study).
* REGISTRATION: Willing to provide tissue, blood, and stool samples for correlative research purposes.
* REGISTRATION: Arm C Only: Negative serology for acute Epstein-Barr virus (EBV) infection (negative EBV viral capsid antigen [VCA] immunoglobulin M [IgM]).

Exclusion Criteria:

* PRE-REGISTRATION: Prior systemic anti-cancer therapy for melanoma (e.g., chemotherapy, hormonal therapy, targeted therapy, immunotherapy including anti-PD-1, anti-PDL1 agents, or other biologic therapies), with the following exceptions: adjuvant treatment with interferon, IL-2, granulocyte-macrophage colony-stimulating factor (GM-CSF) or vaccine therapies are allowed, if discontinued >= 28 days prior to pre-registration.
* PRE-REGISTRATION: Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
* PRE-REGISTRATION: For patients with concurrent diagnosis of primary melanoma with nodal involvement, major surgical procedure other than lymph node biopsy or wide local excision of primary melanoma =< 4 weeks prior to pre-registration, or anticipation of need for a major surgical procedure for reasons other than melanoma during the course of the study.
* PRE-REGISTRATION: For patients with nodal recurrence, surgical procedure or anti-cancer therapy for this recurrence (other than lymph node biopsy) or anticipation of need for a major surgical procedure for reasons other than melanoma during the course of the study.
* PRE-REGISTRATION: Prior radiotherapy for melanoma.
* PRE-REGISTRATION: History of non-nodal melanoma metastasis or central nervous system (CNS) lesion(s) proven or clinically suspected to be metastasis.
* PRE-REGISTRATION: Active malignancy (other than melanoma) or malignancy =< 3 years prior to pre-registration.

  * NOTE: Exceptions: Asymptomatic papillary thyroid cancer (not requiring treatment), resected basal cell carcinoma (BCC), resected cutaneous squamous cell carcinoma (SCC), resected carcinoma in situ of the cervix, resected carcinoma in situ of the breast, in situ prostate cancer, non-muscle-invasive bladder cancer, Stage I uterine cancer, or other curatively treated malignancies from which the patient has been disease-free for at least 3 years prior to pre registration.
* PRE-REGISTRATION: Prior allogeneic stem cell or solid organ transplantation.
* PRE-REGISTRATION: History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* PRE-REGISTRATION: History of autoimmune disease requiring systemic immunosuppressive or immune-modulatory therapy =< 5 years prior to pre-registration.

  * NOTE: Exceptions are allowed for hypothyroidism on thyroid replacement therapy; or Type 1 diabetes on insulin regimen.
* PRE-REGISTRATION: Active psoriasis requiring therapy (systemic or topical).
* PRE-REGISTRATION: Known clinically significant liver disease, including alcoholism, cirrhosis, fatty liver, and other inherited liver disease as well as active viral disease.
* PRE-REGISTRATION: Arms A and B only: History of or evidence of retinal pathology on ophthalmologic examination including but not limited to:

  * Neurosensory retinal detachment
  * Central serous chorioretinopathy
  * Retinal vein occlusion (RVO)
  * Neovascular macular degeneration
* PRE-REGISTRATION: Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* PRE-REGISTRATION: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection (including but not limited to tuberculosis)
  * Clinically significant cardiac dysfunction including:

    * Symptomatic congestive heart failure defined as New York Heart Association class II or higher
    * Unstable angina pectoris or new-onset angina =< 3 months prior to pre-registration
    * Unstable cardiac arrhythmia
    * Myocardial infarction =< 3 months prior to pre-registration
    * Congenital long QT syndrome
  * Clinically significant stroke, reversible ischemic neurological defect, or transient ischemic attack =< 6 months prior to pre-registration
  * Any grade 3 hemorrhage or bleeding event =< 4 weeks prior to pre-registration
  * Uncontrolled diabetes or symptomatic hyperglycemia
  * Psychiatric illness/social situations that, in the judgement of the investigator, would: a) limit compliance with study requirements, or b) make the patient inappropriate for entry into this study, or c) interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* PRE-REGISTRATION: Known hypersensitivity to biopharmaceutical agents produced in Chinese hamster ovary cells (example [ex]: recombinant follicle-stimulating hormone [FSH]).
* PRE-REGISTRATION: Known hypersensitivity to any components of the atezolizumab (all arms), tiragolumab (Arm C only), cobimetinib (Arms A and B only), or vemurafenib (Arms A and B only) formulations.
* PRE-REGISTRATION: History of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* REGISTRATION: Received anticancer treatments or investigational agents during pre-registration period.
* REGISTRATION: Clinically suspected non-nodal metastatic melanoma.
* REGISTRATION: Arm A only: For BRAF-mutant patients only: anticipated use of any concomitant medication =< 7 days prior to registration that is known to cause QT prolongation (which may lead to torsade de pointes).
* REGISTRATION: Arms A and B only: History of malabsorption or other clinically significant metabolic dysfunction that may interfere with absorption of oral study treatment or inability or unwillingness to swallow oral medication.
* REGISTRATION: Signs or symptoms of infection or has received antibiotics =< 14 days prior to registration.

  * NOTE: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* REGISTRATION: Any of the following because this study involves investigational agents whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* REGISTRATION: Treatment with a live, attenuated vaccine =< 4 weeks prior to registration, or anticipation of need for such a vaccine during the course of the study.
* REGISTRATION: Treatment with systemic immunosuppressive medication (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF)-alpha agents) =< 2 weeks prior to registration, or anticipation of need for systemic immunosuppressive medication during the course of the study.

  * NOTE: Patients who have received acute, low-dose systemic steroids (=< 10 mg/day oral prednisone or equivalent) prior to registration or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * NOTE: The use of inhaled corticosteroids for chronic obstructive pulmonary disease or asthma, mineralocorticoids (e.g., fludrocortisone), or low-dose corticosteroids for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* REGISTRATION: Requirement for concomitant therapy or food that is prohibited during the study.
* REGISTRATION: Arms A and B only: Inability to abstain from alcohol during neoadjuvant phase.
* REGISTRATION: Arm C only: Known Epstein-Barr virus (EBV) infection.

  * NOTE: Patients with symptoms such as splenomegaly, fever, sore throat, non-malignant cervical lymphadenopathy, and/or tonsillar exudate, should undergo an EBV polymerase chain reaction (PCR) test to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) in patients with stage III BRAFm (mutant) melanoma (neoadjuvant phase) | After 12 weeks of therapy
  Pathologic complete response rate defined as the percentage of patients with no residual disease found in the surgical specimen among the patients who began neo-adjuvant protocol treatment. An interval estimate will be obtained using the formula for a 90% binomial confidence interval for one sample proportion.
Pathologic complete response rate in patients with stage III BRAFwt (wild type) melanoma (neoadjuvant phase) | After 12 weeks of therapy
  Pathologic complete response rate defined as the percentage of patients with no residual disease found in the surgical specimen among the patients who began neo-adjuvant protocol treatment. An interval estimate will be obtained using the formula for a 90% binomial confidence interval for one sample proportion.
Median recurrence-free (RFS) rate (adjuvant phase) | From surgery assessed up to 3 years
  Recurrence-free survival is defined as the time from surgery to radiographic or histologic evidence of local, regional, or distant recurrence of melanoma or death due to any cause. For each regimen, the distribution of recurrence-free survival times [denoted as RFS(t)] will be estimated using the Kaplan-Meier method. A 90% confidence interval for V(t) = log [-log (RFS(t)] will be constructed and then the inverse transformation exp[-exp v(t)] will be used to obtain a confidence for RFS(t).

SECONDARY OUTCOMES:
Incidence of adverse events per Common Terminology Criteria for Adverse Events (CTCAE) (neoadjuvant phase) | After 12 weeks of therapy
  For each cohort, the frequency and severity of toxicities will be documented using the CTCAE criteria and tabulated for the neo-adjuvant phase and post-operative visit separately.
Change in the uptake on Positron emission tomography (PET)/computed tomography (CT) results | Baseline to end of neo-adjuvant treatment
  For each cohort, the percent change in the uptake on PET/CT scan taken at the completion of neo-adjuvant treatment from that on PET/CT scan taken prior to the start of neo-adjuvant treatment will be determined. Also, the appearance of new sites of uptake in the post neo-adjuvant treatment scan and lack of uptake in the areas where uptake was seen in the pre-treatment scan will be noted.

OTHER OUTCOMES:
Pretreatment soluble (s)PD-L1, pretreatment tumor PD-L1, and pretreatment intracellular Bim in tumor-related T cells | Up to 3 years
  Stratified Cox modeling will be conducted with participant cohort as the strata to obtain a point and interval estimate of the hazard of recurrence among those with biomarker levels thought to be delirious relative to the hazard of recurrence among those with biomarker levels thought not to be delirious.
Molecular features of melanomas and the tumor immune microenvironment evaluated with multiplexed immunohistochemistry (mIHC) and ribonucleic acid sequencing (RNASeq) | Up to 3 years
  Graphs will be constructed to visually compare and contrast the levels of these biomarkers between those who achieve a pCR and those who did not. Binomial confidence intervals for the difference in two independent proportions or t confidence intervals for the difference in two independent means will be used to gain preliminary insights into the difference in these biomarkers among those who achieve a pCR and those who did not.
Changes in the concentration of circulating tumor deoxyribonucleic acid (DNA) during neoadjuvant treatment | Up to 3 years
  Will be correlated with pCR. Graphs will be constructed to visually compare and contrast the level of tumor DNA between those who achieve a pCR and those who do not.
Changes in T cell receptor clonality | Up to 3 years
  A waterfall plot of the percent change will be constructed by pCR status. A two sample Wilcoxon rank sum test will be used to assess whether the percent change in intra-tumoral T cells from the primary lesion or in peripheral blood T cells differ among those who have a pCR and those who do not. Also, the proportion of patients who have a change in intra-tumoral T cell clonality and the proportion of patients who have a change in peripheral blood T cell clonality will be determined. For each of these parameters, a 95% binomial confidence interval for the difference in the parameter between those who have a pCR and those who do not will be constructed. Finally, the ratio of the intra-tumoral T cell clonality in the involved lymph node to the intra-tumoral T cell clonality in the uninvolved lymph node will be determined. This ratio will be summarized descriptively using median and inter-quartile range.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Block, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Result] Hieken TJ, Nelson GD, Flotte TJ, Grewal EP, Chen J, McWilliams RR, Kottschade LA, Yang L, Domingo-Musibay E, Dronca RS, Yan Y, Markovic SN, Dimou A, Montane HN, Erskine CL, Piltin MA, Price DL, Khariwala SS, Hui J, Strand CA, Harrington SM, Suman VJ, Dong H, Block MS. Neoadjuvant cobimetinib and atezolizumab with or without vemurafenib for high-risk operable Stage III melanoma: the Phase II NeoACTIVATE trial. Nat Commun. 2024 Feb 16;15(1):1430. doi: 10.1038/s41467-024-45798-8. PMID 38365756
- [Result] Block MS, Nelson GD, Chen J, Johnson S, Yang L, Flotte TJ, Grewal EP, McWilliams RR, Kottschade LA, Domingo-Musibay E, Markovic SN, Dimou A, Montane HN, Piltin MA, Price DL, Khariwala SS, Hui JYC, Erskine CL, Strand CA, Zahrieh D, Dong H, Hieken TJ. Neoadjuvant cobimetinib and atezolizumab with or without vemurafenib for stage III melanoma: outcomes and the impact of the microbiome from the NeoACTIVATE trial. J Immunother Cancer. 2025 Apr 15;13(4):e011706. doi: 10.1136/jitc-2025-011706. PMID 40234093
- [Result] Hieken TJ, Price DL, Piltin MA, Turner HJ, Block MS. Surgeon Assessment of the Technical Impact of Neoadjuvant Systemic Therapy on Operable Stage III Melanoma. Ann Surg Oncol. 2022 Feb;29(2):780-786. doi: 10.1245/s10434-021-11112-9. Epub 2021 Nov 25. PMID 34825282
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials